CLINICAL TRIAL: NCT06354595
Title: Feasibility Study of Multidimensional Rehabilitation in the Metaverse
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qu Shen (Other)
Collaborators: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor-Investigator, Qu Shen, Associate Professor, Xiamen University
Organization: Xiamen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: XiamenU1
Record Dates: First submitted 2024-03-12; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Colorectal Neoplasms
Keywords: Metaverse multi-dimensional rehabilitation platform
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Colorectal cancer survivors and their families (Other): Using the Colorectal Cancer Survivor Metaverse Multidimensional Rehabilitation Platform, and provide feedback and suggestions.
  Interventions: Device: Multidimensional Rehabilitation in the Metaverse

INTERVENTIONS:
Device: Multidimensional Rehabilitation in the Metaverse — Using the multidimensional rehabilitation space in the metaverse, evaluate the platform after use.

SUMMARY:
The investigators evaluated and optimized the Metaverse multi-dimensional rehabilitation platform based on the use of the Metaverse multi-dimensional rehabilitation platform by colorectal cancer survivors and their families, and finally launched the Metaverse multi-dimensional rehabilitation platform.

DETAILED DESCRIPTION:
The investigatorse intend to invite colorectal cancer survivors and their families to use the metaverse multi-dimensional rehabilitation platform. Interviews with users, user experience optimization of the metaverse multi-dimensional rehabilitation platform, and then evaluation of the platform through system usability evaluation. Gain insight into the experience of colorectal cancer survivors using the metaverse multi-dimensional rehabilitation platform, and understand their opinions and suggestions to explore the usability of the metaverse multi-dimensional rehabilitation platform.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing adjuvant therapy after radical colorectal cancer resection; Age over 18 years old, under 65 years old, non-pregnant; Volunteering to participate in the research of this topic; Mobile phones are available

Exclusion Criteria:

* Patients with multiple cancers; Have special dietary needs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Post-Study System Usability Questionnaire (PSSUQ) Third Edition | 4th week
  The questionnaire includes three dimensions: usefulness, information quality, interface quality, and one overall evaluation item, totaling 20 items. Each item is rated on a scale from 'strongly disagree' to 'strongly agree' with scores ranging from 1 to 5. A higher score indicates higher user satisfaction.
System Usability Scale (SUS) | 4th week
  Used to evaluate user experience, employing the Likert 5-point scale method, consisting of 10 questions. Questions 1, 3, 5, 7, and 9 are positively worded, while questions 2, 4, 6, 8, and 10 are negatively worded. The validity of the scale is 0.85. The SUS is scored on a percentage scale. When the questionnaire score is above 70, the product is considered 'good,' and above 50 is considered 'okay.

SECONDARY OUTCOMES:
Semi-structured interview | 4th week
  Through interviews, conducting interviews with colorectal cancer patients on the theme of 'platform implementation effectiveness' to understand the evaluation of colorectal cancer patients on this mobile healthcare platform.

CONTACTS AND LOCATIONS:
Overall Officials: Yuru HU, Principal Investigator — Xiamen University School of Medicine
Locations (1):
- Yuru Hu, Xiamen, Fujian, China